CLINICAL TRIAL: NCT02371733
Title: Effects of Upper Extremity Aerobic Exercise Training on Functional Exercise Capacity in Patients With Pulmonary Arterial Hypertension
Brief Title: Aerobic Exercise Training in Pulmonary Arterial Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Meral Boşnak Güçlü, Assoc. Prof, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Gazi University2
Record Dates: First submitted 2015-02-20; First posted 2015-02-26 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: pulmonary arterial hypertension; aerobic exercise training; upper extremity; exercise capacity
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Training Group (Active Comparator): Intervention:Training group will receive upper extremity aerobic exercise training using arm ergometer and breathing exercises.
  Interventions: Other: Upper extremity aerobic exercise training
- Control Group (Sham Comparator): Sham: Control group will receive alternative upper extremity exercises and breathing exercises.
  Interventions: Other: Alternative upper extremity exercises

INTERVENTIONS:
Other: Upper extremity aerobic exercise training — Training group will receive upper extremity aerobic exercise training using arm ergometer at 50-80% of maximal heart rate and breathing exercises.
  Training will exercise with arm ergometer 3days/week, for 6 weeks with the assistance of a physiotherapist. Training workload will be undercontrol both using target heart rate and Modified Borg dyspnea scale. Training group will also perform breathing exercises 120 times/day, 7 days/week, for 6 weeks.
  Arms: Training Group
Other: Alternative upper extremity exercises — Control group will receive alternative upper extremity exercises and breathing exercises. Control group will perform alternative upper extremity exercises 3days/week, for 6 weeks and also breathing exercises 120 times/day, 7 days/week, for 6 weeks.
  Control group will be followed-up by telephone once a week.
  Arms: Control Group

SUMMARY:
Decreased exercise capacity, peripheral muscle strength and quality of life and increased dyspnea and fatigue perception is prevalent in patients with pulmonary arterial hypertension. It was demonstrated exercise training has beneficial effects in patients with pulmonary arterial hypertension. However, no study investigated the effects of upper extremity aerobic exercise training, therefore effects of upper extremity aerobic exercise training on outcomes in patients with pulmonary arterial hypertension.

DETAILED DESCRIPTION:
Patients were diagnosed with pulmonary arterial hypertension according to the Task Force for the Diagnosis and Treatment of Pulmonary Hypertension of f the European Society of Cardiology (ESC) and European Respiratory Society (ERS). Primary outcome measurement was exercise capacity, secondary outcomes were respiratory and peripheral muscle strength, physical activity, quality of life, fatigue, dyspnea and depression.

ELIGIBILITY:
Inclusion Criteria:

* Clinically stable
* Under standard medication
* Group 1 pulmonary arterial hypertension patients
* Having no exacerbation or infection

Exclusion Criteria:

* Cognitive disorders
* Orthopedic and neurological problems
* Pneumonia or acute infection
* Stage 4 heart failure
* Having no comorbidity to avoid performing evaluation and training

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-04; Primary Completion 2018-01 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Functional exercise capacity (Oxygen consumption measurement during test) | 6 weeks
  Six minute walk test (6MWT)

SECONDARY OUTCOMES:
Maximum inspiratory and expiratory muscle strength (MIP, MEP) | 6 weeks
  Mouth pressure device
Peripheral muscle strength | 6 weeks
  Hand held dynamometer
Pulmonary functions | 6 week
  Spirometry
Physical activity | 6 weeks
  Activity monitor
Dyspnea | 6 weeks
  Modified Borg and Modified Medical Research Council (MMRC) dyspnea scales
Fatigue | 6 weeks
  Fatigue Severity Scale (FSS)
Generic quality of life | 6 weeks
  Short Form (SF-36) Health Survey
Depression | 6 weeks
  Montgomery Asberg Depression Rating Scale (MADRS) (Turkish versions of all scales)

CONTACTS AND LOCATIONS:
Overall Officials: Burcu Camcıoğlu, MSc, Study Chair — Gazi University; Meral Boşnak Güçlü, PhD, Study Director — Gazi University; Müşerrefe N Karadallı, MSc, Principal Investigator — Gazi University; Gülten Aydoğdu Taçoy, MD, Principal Investigator — Gazi University; Atiye Çengel, MD, Principal Investigator — Gazi University
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

REFERENCES:
- [Result] D'Alonzo GE, Gianotti LA, Pohil RL, Reagle RR, DuRee SL, Fuentes F, Dantzker DR. Comparison of progressive exercise performance of normal subjects and patients with primary pulmonary hypertension. Chest. 1987 Jul;92(1):57-62. doi: 10.1378/chest.92.1.57. PMID 3109813
- [Result] Riley MS, Porszasz J, Engelen MP, Shapiro SM, Brundage BH, Wasserman K. Responses to constant work rate bicycle ergometry exercise in primary pulmonary hypertension: the effect of inhaled nitric oxide. J Am Coll Cardiol. 2000 Aug;36(2):547-56. doi: 10.1016/s0735-1097(00)00727-0. PMID 10933371
- [Result] Deboeck G, Niset G, Lamotte M, Vachiery JL, Naeije R. Exercise testing in pulmonary arterial hypertension and in chronic heart failure. Eur Respir J. 2004 May;23(5):747-51. doi: 10.1183/09031936.04.00111904. PMID 15176691
- [Result] Mereles D, Ehlken N, Kreuscher S, Ghofrani S, Hoeper MM, Halank M, Meyer FJ, Karger G, Buss J, Juenger J, Holzapfel N, Opitz C, Winkler J, Herth FF, Wilkens H, Katus HA, Olschewski H, Grunig E. Exercise and respiratory training improve exercise capacity and quality of life in patients with severe chronic pulmonary hypertension. Circulation. 2006 Oct 3;114(14):1482-9. doi: 10.1161/CIRCULATIONAHA.106.618397. Epub 2006 Sep 18. PMID 16982941
- [Result] McKeough ZJ, Bye PT, Alison JA. Arm exercise training in chronic obstructive pulmonary disease: a randomised controlled trial. Chron Respir Dis. 2012 Aug;9(3):153-62. doi: 10.1177/1479972312440814. Epub 2012 Mar 27. PMID 22452973
- [Result] Nyquist-Battie C, Fletcher GF, Fletcher B, Carlson JM, Castello R, Oken K. Upper-extremity exercise training in heart failure. J Cardiopulm Rehabil Prev. 2007 Jan-Feb;27(1):42-5. doi: 10.1097/01.hcr.0000265019.18661.82. PMID 17474643
- [Derived] Yilmaz BC, Guclu MB, Keles MN, Tacoy GA, Cengel A. Effects of upper extremity aerobic exercise training on oxygen consumption, exercise capacity, dyspnea and quality of life in patients with pulmonary arterial hypertension. Heart Lung. 2020 Sep-Oct;49(5):564-571. doi: 10.1016/j.hrtlng.2020.04.006. Epub 2020 May 24. PMID 32457004